CLINICAL TRIAL: NCT01786408
Title: A Study to Compare Analyte Levels in Blood Samples Collected Using the TAP20-C Device With Results Obtained by Fingerstick Using the SAFE-T-FILL Capillary Blood Collection System
Brief Title: A Study to Compare Analytes in Blood Collected Using an Investigational Collection Device With a Commercial Predicate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Seventh Sense Biosystems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-P001
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Last update posted 2014-11-25 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes; Anemia
MeSH Terms: conditions — Diabetes Mellitus; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAP20-C (Experimental): Single Use Integrated Capillary Blood Collection System
  Interventions: Device: TAP20-C
- SAFE-T-FILL CAPILLARY SYSTEM (Active Comparator): Single Use Capillary Blood Collection System
  Interventions: Device: SAFE-T-FILL CAPILLARY BLOOD COLLECTION SYSTEM

INTERVENTIONS:
Device: TAP20-C
  Arms: TAP20-C
Device: SAFE-T-FILL CAPILLARY BLOOD COLLECTION SYSTEM
  Arms: SAFE-T-FILL CAPILLARY SYSTEM

SUMMARY:
This study will involve an investigational device, the Seventh Sense Biosystems TAP20-C. The TAP20-C device collects small amounts of blood from the forearm which can then be used for blood testing. The study will also involve collecting blood by fingerstick which is a common way of collecting blood. The SAFE-T-FILL Capillary Blood Collection system and the Terumo Capiject 1.5 mm Blade Safety Lancet will be used for this. The study will compare the concentrations of glucose, hemoglobin, and HbA1C in blood samples collected with the two different blood collection methods. Additional information will be collected about how the TAP20-C device performs.

ELIGIBILITY:
Inclusion Criteria:

Healthy Subject Group

1. Male and female volunteers 18 years of age or older

Diabetic Subject Group

1. Male and female volunteers 18 years of age or older
2. Have been diagnosed with Type 1 or Type 2 diabetes mellitus by self-report

Exclusion Criteria:

1.Subjects who are pregnant or nursing mothers by self report 2.Subjects who have eaten or consumed sugar-containing drinks in the 2 hours before blood sample collection begins 3.Subjects with a history of skin disorders or who present with abnormal skin integrity or atypical skin health within the areas to be tested 4.Subjects with a missing index or middle finger on either hand or a missing forearm 5.Subjects who have known allergies to titanium

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Non-Inferiority of Analyte Levels | Day 1
  The study will compare the concentrations of glucose, hemoglobin, and HbA1C in blood samples collected with the two different blood collection methods in a single two hour session.

CONTACTS AND LOCATIONS:
Locations (1):
- Seventh Sense BIosystems, Cambridge, Massachusetts, United States